CLINICAL TRIAL: NCT02748096
Title: The Assessment of Patient Specific Instrumentation for Unicompartmental Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7110
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2016-04

CONDITIONS: Knee Arthritis
Keywords: Unicompartmental Knee Replacement; Patient Specific Instrumentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Specific Instrumentation (Experimental): Patients undergoing unicompartmental knee replacement with the additional aid of patient specific instrumentation.
  Interventions: Procedure: Patient Specific Instrumentation
- Conventional Instrumentation (Active Comparator): Patients undergoing unicompartmental knee replacement using standard instrumentation.
  Interventions: Procedure: Conventional Instrumentation

INTERVENTIONS:
Procedure: Patient Specific Instrumentation — Patients will undergo a medial unicompartmental knee replacement. This knee replacement is implanted using patient specific cutting guides that have been produced based on the patient's individual anatomy (using plans from pre-operative MRI scans of the patient's knee).
  Arms: Patient Specific Instrumentation
Procedure: Conventional Instrumentation — Patients will undergo a medial unicompartmental knee replacement using standard conventional instruments.
  Arms: Conventional Instrumentation

SUMMARY:
Patient-specific instrumentation guides have previously been used to improving surgical accuracy and ease of implantation during Total Knee Replacement but have received less attention for implanting Unicompartmental Knee Replacement. The aim of this prospective study is to compare the accuracy of implantation and functional outcome of mobile bearing medial Unicompartmental Knee Replacement implanted with and without patient specific instrumentation by experienced knee surgeons.

DETAILED DESCRIPTION:
The aim of this prospective study is to compare the accuracy of implantation and functional outcome of mobile bearing medial Unicompartmental Knee Replacements implanted with and without patient specific instrumentation by experienced Unicompartmental Knee Replacement surgeons.

This single-centre parallel-design trial was conducted between March 2012 and March 2014 at the Nuffield Orthopaedic Centre, Oxford. Four expert knee surgeons performed all of the procedures in this study. Patients who were being placed on the waiting list for a medial Unicompartmental Knee Replacement, and met the entry criteria for the trial, were asked to see if they would be willing to receive further information about participation in the study. They were provided with a study information leaflet that they could read in their own time. A member of the research team subsequently contacted the patients in order to determine if they would agree to take part in the study and enrolled them onto the study.

Patients were randomized to either Patient Specific Instrumentation, or Conventional Instrumentation group. There were 23 patients (23 knees) in the Patient Specific Instrumentation group and 22 patients (22 knees) in the Conventional Instrumentation group. Randomization was performed using sealed opaque envelopes. Concealment from operating surgeons and patients was not possible owing to the surgeon needing to confirm the Patient Specific Instrumentation plans, and the patients undergoing pre-operative MRI scans. Patient Specific Instrumentation group patients underwent an MRI scan using the protocol outlined by the Patient Specific Instrumentation manufacturers to plan development of the Patient Specific Instrumentation guides. The preliminary plan indicating prosthesis size, positioning, alignment, and proposed bone resection levels was reviewed by the surgeons who accepted the default preoperative plans unless gross errors were present. The patient specific cutting blocks were then manufactured and sent for sterilization.

Operative Technique:

All patients received a mobile bearing medial Oxford unicompartmental knee replacement via a minimally invasive approach under general anaesthetic, and high thigh tourniquet. Intra-operatively, the bone cuts were made through the Patient Specific Instrumentation guides without the use of any intra or extra-medullary instrumentation on the femoral side but with a tibial extramedullary guide for some cases. The subsequent milling process and all soft tissue balancing was performed manually in the standard fashion.

Post-operatively, the need to have a blood transfusion, and the change haemoglobin levels were also recorded. Oxygen saturation levels over the first 24 hours post surgery were also recorded. Screened anteroposterior and lateral post-operative radiographs were performed prior to discharge. Patients attended the physiotherapy ward discharge clinic at six weeks. A further clinical review was performed at 12 months at which point Oxford Knee Scores were recorded.

The primary outcome measure was radiological assessment of component positioning. (See Outcome measures section for more detail)

Target sample size:

The sample size was calculated from a previous study that used similar radiological assessments to compare unicompartmental knee replacements performed using conventional instrumentation, with those performed using computer navigation. In this study, the standard deviation of the tibia varus/valgus angle for the control group was 3.6°. Assuming a minimum clinically important difference of 3°, the standard mean difference would be 0.8. Hence with a power of 0.8 and significance level of 0.05, a total sample size of 44 patients (22 in each group) was required.

ELIGIBILITY:
Inclusion Criteria:

* Both cruciate ligaments functionally intact
* Full thickness cartilage in the lateral compartment
* Correctable intra-articular varus deformity
* Full thickness cartilage loss in the medial compartment

Exclusion Criteria:

* Contra-indication for MRI
* All forms of inflammatory arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Price, FRCS PhD, Principal Investigator — Nuffield Department of Orthopaedics, Rheumatology & Musculoskeletal Sciences, University of Oxford

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish in high impact peer reviewed orthopaedic journal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.80 (7.17) | 68.18 (10.40) | 67.50 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Radiological Assessment of Component Positioning
Description: Radiological assessment of component positioning and alignment based on post-operative knee radiographs.
Time Frame: Within a weeks after surgery
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Number analyzed (Participants) | 23 | 22
Degrees
  Femur: varus/valgus angle | 0.9 (4.0) | 1.8 (3.0)
  Femur: flexion/extension angle | 9.1 (3.0) | 8.8 (4.8)
  Tibia: varus/valgus angle | 3.5 (2.9) | 8.8 (4.8)
  Tibia:posterior tilt angle | 3.5 (2.9) | 4 (2.1)
  Tibia: posterior tilt angle | 1.8 (2.8) | 3.7 (2.1)
  Tibia: medial fit | 0 (1.0) | 1.0 (1.3)
  Tibia: anterior fit | 1.0 (0.9) | 1.0 (0.7)
  Tibia: posterior fit | 0 (0.8) | 0 (0.9)
Statistical Analysis 1: Comparison: Patient Specific Instrumentation vs Conventional Instrumentation; The sample size was calculated from a previous study that used similar radiological assessments to compare OUKAs performed using conventional instrumentation and computer navigation. In this study, the standard deviation of the tibia varus/valgus angle for the control group was 3.6°. Assuming a minimum clinically important difference of 3°, the SMD would be 0.8. Hence with a power of 0.8 and significance level of 0.05, a total sample size of 44 patients (22 in each group) was required; Test type: Other; p < 0.05, t-test, 2 sided — A p value of less than 0.05 was considered statistically significant for all the radiographic parameters; This test applies to comparison between the two treatment arms and assesses all the radiographic parameters

2. Secondary Outcome: Assessment of Functional Outcome
Description: Use of the patient reported outcome tool (Oxford Knee Score) to determine functional outcome at one year following surgery.
  Total score is 48. Minimum score 0 and Maximum score 48 with higher score indicating better function.
  Scores on a scale
Time Frame: One year after surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Number analyzed (Participants) | 23 | 22
score on a scale | 18.3 [4 to 31] | 18.2 [5 to 31]
Statistical Analysis 1: Comparison: Patient Specific Instrumentation vs Conventional Instrumentation; Test type: Other; p < 0.05, t-test, 2 sided

3. Other Pre Specified Outcome: Post-operative Change in Haemoglobin Between Baseline Baseline and 48 Hours After Surgery
Description: Change in haemoglobin levels between baseline and 48 hours after surgery will be determined
Time Frame: Within the first 48 hours after surgery
Population: Mean drop in post-operative Haemoglobin
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Number analyzed (Participants) | 23 | 22
g/dl | 1.66 (0.79) | 1.80 (0.59)
Statistical Analysis 1: Comparison: Patient Specific Instrumentation vs Conventional Instrumentation; Test type: Other; p < 0.05, t-test, 2 sided

4. Other Pre Specified Outcome: Number of Participants With The Need for Blood Transfusion Following Surgery
Description: Number of Participants with The Need for Blood Transfusion within 48 hours of Surgery
Time Frame: Within the first 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Number analyzed (Participants) | 23 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Patient Specific Instrumentation | Conventional Instrumentation
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Specific Instrumentation (N=23) | Conventional Instrumentation (N=22)
Superficial wound infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — There were two superficial wound infections (one in each group), which were treated by the patients' family physicians which were treated with oral antibiotics and fully resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes